CLINICAL TRIAL: NCT02076425
Title: A Randomized Controlled Trial of PCIT-ED for Preschool Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH098454-02 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Child Psychiatry; Parent-Child Relationship; Therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCIT-ED (Experimental): Parent-Child Interaction Therapy - Emotional Development (PCIT-ED) is a promising early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention.
  Interventions: Behavioral: PCIT-ED
- Wait List (No Intervention): No intervention while subjects wait for PCIT-ED in the second phase of the study.

INTERVENTIONS:
Behavioral: PCIT-ED
  Arms: PCIT-ED

SUMMARY:
Parent Child Interaction Therapy Emotion Development (PCIT-ED) will be conducted with a sample of preschoolers who exhibit symptoms of depression compared to a wait list (WL) control after which participants will receive the active treatment. PCIT-ED is an expansion of PCIT, a well-known, widely used and proven effective treatment for preschool disruptive disorders. To address early disturbances of mood and affect, a novel ED module was added based on empirical data in emotion development. The ED module targets parent emotion learning skills with the goal of training the parent to serve as a more effective emotion teacher and coach to the child. The goal of the ED module is to enhance the child's capacity for emotion recognition and regulation or "emotional competence." In order to test the efficacy of PCIT-ED, to estimate accurate effect sizes and to investigate mediators and moderators of treatment response participants will complete comprehensive pre-, interval, and post-assessments.

Preschoolers over 3 will be offered the option of enrolling in an add-on electroencephalography and magnetic resonance imagery study, to investigate neural changes associated with PCIT-ED.

Compared to those randomized to the WL, preschoolers who undergo PCIT-ED will show significantly increased rates of remission, greater reductions in MDD symptoms, and decreases in impairment; and will show significantly greater increases in emotional competence measured by the ability to accurately identify emotions in themselves and others and the ability to effectively regulate intense emotions. Compared to those on the WL, parents who undergo PCIT-ED will show significantly greater increases in emotion skill learning and reductions in MDD symptoms and parenting stress.

ELIGIBILITY:
Inclusion Criteria:

* Children who meet all DSM-IV MDD symptom criteria (adjusted for development)

Exclusion Criteria:

* Children with serious chronic medical illness
* Children with Autistic Spectrum Disorders (based on clinical diagnosis or Social Responsiveness Scale scores which will be administered when there is suspicion of an ASD)
* Children with significant speech delays
* Children with general developmental delays or IQ < 70
* Children with chronic neurological problems/illnesses
* Children adopted after 12 months of age
* Children on antidepressants
* Children taking unstable doses of other psychotropic medications without antidepressant properties
* Children participating in ongoing psychotherapy
* Children in unstable placements (not with same caregiver for 6 months prior to study enrollment)
* Children who are too ill to wait 18 weeks for treatment (e.g. having active suicidal ideation and/or in acute/serious distress)

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Luby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Early Emotional Development Program, St Louis, Missouri, United States

REFERENCES:
- [Background] Luby J, Lenze S, Tillman R. A novel early intervention for preschool depression: findings from a pilot randomized controlled trial. J Child Psychol Psychiatry. 2012 Mar;53(3):313-22. doi: 10.1111/j.1469-7610.2011.02483.x. Epub 2011 Oct 31. PMID 22040016
- [Result] Luby JL, Barch DM, Whalen D, Tillman R, Freedland KE. A Randomized Controlled Trial of Parent-Child Psychotherapy Targeting Emotion Development for Early Childhood Depression. Am J Psychiatry. 2018 Nov 1;175(11):1102-1110. doi: 10.1176/appi.ajp.2018.18030321. Epub 2018 Jun 20. PMID 29921144
- [Result] Luby JL, Gilbert K, Whalen D, Tillman R, Barch DM. The Differential Contribution of the Components of Parent-Child Interaction Therapy Emotion Development for Treatment of Preschool Depression. J Am Acad Child Adolesc Psychiatry. 2020 Jul;59(7):868-879. doi: 10.1016/j.jaac.2019.07.937. Epub 2019 Jul 31. PMID 31376501
- [Result] Barch DM, Whalen D, Gilbert K, Kelly D, Kappenman ES, Hajcak G, Luby JL. Neural Indicators of Anhedonia: Predictors and Mechanisms of Treatment Change in a Randomized Clinical Trial in Early Childhood Depression. Biol Psychiatry. 2019 May 15;85(10):863-871. doi: 10.1016/j.biopsych.2018.11.021. Epub 2018 Dec 4. PMID 30583852 (Retraction: PMID 33153528 Biol Psychiatry. 2020 Dec 1;88(11):888)
- [Derived] Schwartz KTG, Chronis-Tuscano A, Tillman R, Whalen D, Gilbert KE, Luby J. Parent-child psychotherapy targeting emotion development: unpacking the impact of parental depression on child, parenting and engagement outcomes. Eur Child Adolesc Psychiatry. 2023 Dec;32(12):2491-2501. doi: 10.1007/s00787-022-02093-5. Epub 2022 Oct 10. PMID 36216984
- [Derived] Donohue MR, Hoyniak CP, Tillman R, Barch DM, Luby J. Callous-Unemotional Traits as an Intervention Target and Moderator of Parent-Child Interaction Therapy-Emotion Development Treatment for Preschool Depression and Conduct Problems. J Am Acad Child Adolesc Psychiatry. 2021 Nov;60(11):1394-1403. doi: 10.1016/j.jaac.2021.03.018. Epub 2021 May 20. PMID 33865929
- [Derived] Barch DM, Whalen D, Gilbert K, Kelly D, Kappenman ES, Hajcak G, Luby JL. Neural Indicators of Anhedonia: Predictors and Mechanisms of Treatment Change in a Randomized Clinical Trial in Early Childhood Depression. Biol Psychiatry. 2020 Dec 1;88(11):879-887. doi: 10.1016/j.biopsych.2020.06.032. PMID 33153527
- [Derived] Hoyniak CP, Whalen DJ, Barch D, Luby JL. Sleep problems in preschool-onset major depressive disorder: the effect of treatment with parent-child interaction therapy-emotion development. Eur Child Adolesc Psychiatry. 2021 Sep;30(9):1463-1474. doi: 10.1007/s00787-020-01641-1. Epub 2020 Sep 15. PMID 32935261
- [Derived] Whalen DJ, Gilbert KE, Luby JL. Changes in self-reported and observed parenting following a randomized control trial of parent-child interaction therapy for the treatment of preschool depression. J Child Psychol Psychiatry. 2021 Jan;62(1):86-96. doi: 10.1111/jcpp.13263. Epub 2020 May 29. PMID 32469454
- [Derived] Whalen DJ, Gilbert KE, Kelly D, Hajcak G, Kappenman ES, Luby JL, Barch DM. Preschool-Onset Major Depressive Disorder is Characterized by Electrocortical Deficits in Processing Pleasant Emotional Pictures. J Abnorm Child Psychol. 2020 Jan;48(1):91-108. doi: 10.1007/s10802-019-00585-8. PMID 31515716
- [Derived] Gilbert K, Barch DM, Luby JL. The Overcontrol in Youth Checklist (OCYC): Behavioral and Neural Validation of a Parent-Report of Child Overcontrol in Early Childhood. Child Psychiatry Hum Dev. 2020 Feb;51(1):27-38. doi: 10.1007/s10578-019-00907-3. PMID 31256293
- [Derived] Luby JL, Whalen D, Tillman R, Barch DM. Clinical and Psychosocial Characteristics of Young Children With Suicidal Ideation, Behaviors, and Nonsuicidal Self-Injurious Behaviors. J Am Acad Child Adolesc Psychiatry. 2019 Jan;58(1):117-127. doi: 10.1016/j.jaac.2018.06.031. Epub 2018 Oct 22. PMID 30577927
- [Derived] Belden AC, Irvin K, Hajcak G, Kappenman ES, Kelly D, Karlow S, Luby JL, Barch DM. Neural Correlates of Reward Processing in Depressed and Healthy Preschool-Age Children. J Am Acad Child Adolesc Psychiatry. 2016 Dec;55(12):1081-1089. doi: 10.1016/j.jaac.2016.09.503. Epub 2016 Oct 4. PMID 27871643
- See also: Early Emotional Development Program Website — http://eedp.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- PCIT-ED: Parent-Child Interaction Therapy - Emotional Development (PCIT-ED) is a promising early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention.
  PCIT-ED
Period: Overall Study
Arm/Group | PCIT-ED | Wait List
Started | 114 | 115
Completed | 100 | 91
Not Completed | 14 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCIT-ED | Wait List | Total
Number analyzed (Participants) | 114 | 115 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.14 (0.97) | 5.28 (1.13) | 5.21 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 76 | 73 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 99 | 105 | 204
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 18 | 27
  White | 94 | 82 | 176
  More than one race | 10 | 15 | 25
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 115 | 229
K-SADS-EC MDD Core Symptom Score [Mean (Standard Deviation); unit: units on a scale] — The Kiddie Schedule for Affective Disorders and Schizophrenia - Early Childhood (K-SADS-EC) is a semi-structured clinical interview for DSM-5 disorders adapted for use in children aged 3-6. The MDD core symptom score was the number of core MDD symptoms endorsed on the K-SADS-EC. These 9 symptoms were (1) depressed mood, (2) anhedonia, (3) insomnia/hypersomnia, (4) fatigue, (5) decreased concentration, (6) weight/appetite change, (7) psychomotor agitation/retardation, (8) worthlessness/guilt, (9) suicidal thoughts/behaviors. The range of possible values is 0-9, with 9 being the worst outcome.
  units on a scale | 5.49 (1.47) | 5.71 (1.51) | 5.60 (1.49)
Preschool Feelings Checklist-Scale Version (PFC-Scale) Score [Mean (Standard Deviation); unit: units on a scale] — The Preschool Feelings Checklist - Scale Version (PFC-Scale), was adapted from the PFC, which is a validated screening checklist used to capture young children at high risk for MDD. The PFC-Scale is a 23-item Likert scale with possible values of 0, 1, 2, 3, or 4 for each item. The total score is a sum of the 23 items, so the range of possible values is 0-92, with 92 being the most severe score possible.
  units on a scale | 38.77 (9.57) | 41.71 (11.37) | 40.25 (10.59)
Children's Global Assessment Scale (CGAS) Score [Mean (Standard Deviation); unit: units on a scale (0-100)] — The Children's Global Assessment Scale (CGAS) is a standardized instrument that measures children's global level of impairment completed by the clinician-rater. The possible range of values is 0-100, with 0 indicating the most severe global impairment.
  units on a scale (0-100) | 44.00 (6.51) | 42.61 (6.57) | 43.30 (6.56)

OUTCOME MEASURES:

1. Primary Outcome: Kiddie Schedule for Affective Disorders and Schizophrenia - Early Childhood (KSADS-EC) MDD Core Symptom Score
Description: The Kiddie Schedule for Affective Disorders and Schizophrenia - Early Childhood (K-SADS-EC) is a semi-structured clinical interview for DSM-5 disorders adapted for use in children aged 3-6. The MDD core symptom score was the number of core MDD symptoms endorsed on the K-SADS-EC. These 9 symptoms were (1) depressed mood, (2) anhedonia, (3) insomnia/hypersomnia, (4) fatigue, (5) decreased concentration, (6) weight/appetite change, (7) psychomotor agitation/retardation, (8) worthlessness/guilt, (9) suicidal thoughts/behaviors. The range of possible values is 0-9, with 9 being the worst outcome.
Time Frame: completion of therapy (average of 20 weeks)
Measure: Mean (Standard Deviation); unit: number of symptoms (0-9)
Arm/Group | PCIT-ED | Wait List
Number analyzed (Participants) | 100 | 91
number of symptoms (0-9) | 1.74 (1.69) | 4.15 (2.04)

2. Secondary Outcome: Preschool Feelings Checklist-Scale Version (PFC-Scale) Score
Description: The Preschool Feelings Checklist - Scale Version (PFC-Scale), was adapted from the PFC, which is a validated screening checklist used to capture young children at high risk for MDD. The PFC-Scale is a 23-item Likert scale with possible values of 0, 1, 2, 3, or 4 for each item. The total score is a sum of the 23 items, so the range of possible values is 0-92, with 92 being the most severe score possible.
Time Frame: completion of therapy (average of 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCIT-ED | Wait List
Number analyzed (Participants) | 99 | 90
units on a scale | 20.13 (9.68) | 33.24 (11.12)

3. Other Pre Specified Outcome: Children's Global Assessment Scale (CGAS) Score
Description: The Children's Global Assessment Scale (CGAS) is a standardized instrument that measures children's global level of impairment completed by the clinician-rater. The possible range of values is 0-100, with 0 indicating the most severe global impairment.
Time Frame: completion of therapy (average of 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | PCIT-ED | Wait List
Number analyzed (Participants) | 100 | 91
units on a scale (0-100) | 76.83 (16.61) | 55.75 (17.14)

ADVERSE EVENTS:
Time Frame: Baseline assessment through study completion (approximately 40 weeks)
Arm/Group | PCIT-ED | Wait List
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/115
Other Adverse Events (participants affected / at risk) | 0/114 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02076425/Prot_SAP_000.pdf